CLINICAL TRIAL: NCT05104125
Title: A Phase II Randomized, Double-blind, Placebo-controlled, Multi-center, Multi-dose Study to Evaluate Safety and Efficacy of ASC40 Tablets in Subjects With Moderate to Severe Acne Vulgaris.
Brief Title: Study to Evaluate the Safety and Efficacy of ASC40 in Subjects With Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC40-202
Record Dates: First submitted 2021-10-26; First posted 2021-11-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2023-05

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; ASC40
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental group 1 (Experimental): ASC40 25mg for 12 weeks
  Interventions: Drug: ASC40 25mg
- Experimental group 2 (Experimental): ASC40 50mg for 12 weeks
  Interventions: Drug: ASC40 50mg
- Experimental group 3 (Experimental): ASC40 75mg for 12 weeks
  Interventions: Drug: ASC40 75mg
- Placebo group (Placebo Comparator): Placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASC40 25mg — 25mg of ASC40 orally once daily for 12 weeks.
  Arms: Experimental group 1
Drug: ASC40 50mg — 50mg of ASC40 orally once daily for 12 weeks.
  Arms: Experimental group 2
Drug: ASC40 75mg — 75mg of ASC40 orally once daily for 12 weeks.
  Arms: Experimental group 3
Drug: Placebo — Placebo orally once daily for 12 weeks.
  Arms: Placebo group

SUMMARY:
This is a phase2, randomized, double-blind, multi-center, multi-dose and placebo parallel controlled design. The subjects in the study group were given double-blind drugs, and they were taken (orally) after dinner every day according to the requirements of clinical trial scheme.

ELIGIBILITY:
Key Inclusion Criteria:

* 18-40 years old (including 18 and 40 years old);
* Investigator's Global Assessment of subject at baseline period was at 3-4.
* Facial skin lesions of subject need counting as follows: 30 ~ 75 inflammatory lesions (the total number of papules, pustules and nodules is 30 ~ 75, including no more than 2 nodules), 30 ~ 100 non-inflammatory lesions (the total number of open and closed comedones is 30 ~ 100);

Key Exclusion Criteria:

* Known to be allergic or hypersensitive to ASC40 tablets;
* Facial nodules of subject is more than 2 facial nodules
* The subject with cystic acne
* Subject with secondary acne such as occupational acne (e.g., chloroacne) and acne caused by corticosteroids (e.g., chloroacne or acne caused by drugs);
* Serum AST, ALT≥3ULN and Cr exceeded the upper limit of normal range

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Percentage change of total lesion count compared with baseline and week 12. | Baseline to week 12
Ratio of subjects, whose IGA grades was decreased by ≥2 grades compared with baseline at week 12. | Baseline to week 12

SECONDARY OUTCOMES:
The changes status and changes of average percentage of inflammatory skin lesions count, non-inflammatory skin lesions count and total skin lesions count compared with baseline. | Baseline to week 2, 4, 8 and 12
Ratio of subjects, whose GA grades was 1 or 0, or GA grades was decreased y ≥2 grades compared with baseline and Improvements in classification | Baseline to week 2, 4, 8 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen Q, Chen R, Wu L, Xu A, He L, Wang J, Lu Y, Xiao R, Liu L, Feng Y, Zhang C, Dai X, Gao Y, Yan Y, Wu JJ, Xiang L. Denifanstat for moderate-to-severe acne: A Phase 2, randomized, double-blind, placebo-controlled trial. J Eur Acad Dermatol Venereol. 2025 Nov 4. doi: 10.1111/jdv.70119. Online ahead of print. PMID 41186280